CLINICAL TRIAL: NCT06788119
Title: Analyzing the Benefits of Using SYMPTOMS-JIT for in Vivo Exposure in Anxiety Disorders: a Randomized Controlled Trial Using a Mixed Methods Approach
Brief Title: Analyzing the Benefits of Using SYMPTOMS-JIT for in Vivo Exposure in Anxiety Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJaumeI_Symptoms_1
Record Dates: First submitted 2024-12-19; First posted 2025-01-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Anxiety Disorders; Specific Phobia; Panic Disorder; Agoraphobia; Social Anxiety Disorder
Keywords: Anxiety disorders; In vivo exposure; app; smartphone; smartwatch
MeSH Terms: conditions — Anxiety Disorders; Phobia, Specific; Panic Disorder; Agoraphobia; Phobia, Social; Alzheimer Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT Treatment with in vivo exposure (Active Comparator): In this condition participants will receive CBT treatment and be exposed to in vivo situations.
  Interventions: Behavioral: Cognitive behavioral therapy with in vivo exposure
- CBT Treatment with in vivo exposure plus SYMPTOMS-JIT (Experimental): In this condition participants will receive CBT treatment and be exposed to in vivo situations with the support of SYMPTOMS-JIT.
  Interventions: Behavioral: Cognitive behavorial therapy with in vivo exposure plus SYMPTOMS-JIT

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy with in vivo exposure — CBT will be used as the chosen approach for ADs. The main components will be psychoeducation and to help patients to challenge and change unhelpful cognitive distortions (e.g., thoughts, beliefs, and attitudes) and behaviors (e.g., avoidance), develop emotion regulation strategies (e.g., cognitive reappraisal), and learn coping strategies that target problem-solving. The practice is developed in several sessions that usually last between 10 and 20 sessions. Specifically, the exposure component will be considered as the first-line treatment. During the exposure component, patients will confront themselves over a long period of time, repetitively, with a feared stimulus until distress has decreased significantly by the exposure.In this condition participants will receive CBT treatment and be exposed to in vivo situations.
  Arms: CBT Treatment with in vivo exposure
Behavioral: Cognitive behavorial therapy with in vivo exposure plus SYMPTOMS-JIT — CBT will be used as the chosen approach for ADs. The main components will be psychoeducation and to help patients to challenge and change unhelpful cognitive distortions (e.g., thoughts, beliefs, and attitudes) and behaviors (e.g., avoidance), develop emotion regulation strategies (e.g., cognitive reappraisal), and learn coping strategies that target problem-solving. The practice is developed in several sessions that usually last between 10 and 20 sessions. Specifically, the exposure component will be considered as the first-line treatment. During the exposure component, patients will confront themselves over a long period of time, repetitively, with a feared stimulus until distress has decreased significantly by the exposure. In this condition participants will receive CBT treatment and be exposed to in vivo situations with the support of SYMPTOMS-JIT.
  Arms: CBT Treatment with in vivo exposure plus SYMPTOMS-JIT

SUMMARY:
The aim of this study is to develop and test the efficacy of first-of-its-kind, fully instrumented sensor-based smartphone-guided in-vivo exposure therapy using a just-in-time intervention for anxiety disorder. The main hypotheses are:

1. Both treatment conditions (CBT treatment with IVE and CBT treatment with IVE+SYMPTOMS-JIT) will show efficacy and no statistically significant differences will be found between them. The efficacy will be determined for the differences in pre-post treatment in the used outcome measures.
2. The therapeutic gains obtained in both treatment conditions (IVE and (IVE+SYMPTOMS-JIT) will be maintained at 1-, 6-, and 12-month follow-up periods.
3. Both treatment conditions will be efficient, that is, they will be well-valued by patients and therapists. However, IVE+SYMPTOMS-JIT will be preferred and perceived as less aversive than IVE.
4. The main barriers for the use of this technology are not technological, but rather attitudinal and they can be identified through qualitative studies.

DETAILED DESCRIPTION:
Anxiety Disorders are one of the most prevalent psychological problems around the world and if not treated they tend to become chronic. Cognitive Behavioral Therapy (CBT) is the treatment of choice, being the component of in vivo exposure (IVE) the central feature. Despite its efficacy it is still a hard component to implement for the patients. Information and Communication Technologies (ICT) can help assisting and/or applying psychological interventions. The proposed study will fill the existing gap in this sense as it will assess the efficacy of a fully configurable, sensor-guided and location-based (GPS) app for the in vivo exposure component. It will also address the shortage of clinical validation studies of mHealth apps thanks to the proposed RCT. The study will expand our knowledge about the use of technologies in mental health problems and help improve the effectiveness of exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years or older.
* Meeting DSM-5 diagnostic criteria (APA, 2013) for anxiety disorder, specifically specific phobia, agoraphobia, panic disorder and social phobia.
* Being willing to follow the study conditions.
* Sign the consent form.

Exclusion Criteria:

* Having another psychological problem that requires immediate attention.
* Having current alcohol or drug dependence or abuse, psychosis or severe organic illness.
* Currently being treated in a similar treatment program.
* Taking anxiolytics during the study (or in the case of taking them, changing drug or dose during the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV-TR (ADIS-IV) | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  It is a specific diagnostic semistructured interview for the diagnosis of anxiety disorders. Phobias, Agoraphobia and Social Phobia Sections will be used. For the majority of anxiety disorders, this interview has demonstrated appropriate psychometric qualities and good to exceptional reliability (Orsillo & Roemer, 2001). This instrument includes relevant clinical measures such as interference and distress as perceived by the participant on a scale from 0 to 8 (wherein 0 = "Not at all" and 8 = "Very severe")
Fear and avoidance scales | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The participants and therapists identify the situations and physical sensations that cause the participants the most fear and distress, as well as the negative thoughts associated with them. Next, they assess, on a scale of 0-10, the degree of fear (0="no fear"; 10="extreme fear") and avoidance (0="never avoid"; 10="always avoid") for each feared situation and sensation. In addition, the degree of belief in the negative thoughts related with the target behaviors and sensations are also assessed, using a scale ranging from 0 ("I do not believe the content of the thought at all") to 10 ("I believe the thought is totally true")

SECONDARY OUTCOMES:
Severity Measure for Specific Phobia - Adult | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The SMSP-A is a 10-item measure that assesses the severity of specific phobia in adults during the last 7 days. Each item is rated on a 5-point scale, from 0 (never) to 4 (all of the time). Greater scores indicate more severe specific phobia, being the overall score 40.
Acrophobia Questionnaire | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The AQ evaluates severity of anxiety and avoidance related to different situations that have to do with heights. It consists of 40 items divided into two subscales. On the one hand, there is an anxiety subscale where it is necessary to indicate the degree of anxiety, tension, or discomfort caused in the situations described, responding on a 0 to 6 point Likert-type scale ("no anxiety, calm and relaxed" - "extremely anxious"); and on the other hand, there is an avoidance subscale, where the response is coded on a 0 to 2 point Likert-type scale ("I would not try to avoid it" - "I would not bear it under any circumstances")
Claustrophoby Questionnaire | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The CLQ consists of descriptions of 26 claustrophobic situations. Participants are asked about the degree to which they would feel anxious in these situations according to a 5-alternative Likert-type scale, where (0) is "not at all anxious" and (4) is "extremely anxious." The CLQ consists of two subscales: restriction of movement, ranging from items 1 to 12, and suffocation, ranging from items 13 to 26.
Fear of Flying Questionnaire II | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  This is a list of 30 situations related to flying that can cause discomfort or anxiety, divided into three subscales: in-flight situations, pre-flight situations, and vicarious situations. The items (each representing a situation) are rated on Likert scales from 1 (minimal discomfort) to 10 (maximum discomfort), and therefore the score ranges from 30 to 300.
Anxiety Sensitivity Inventory | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The ASI is a scale composed of 16 items specifying a possible negative consequence to anxiety: additional anxiety or fear, illness, embarrassment and loss of control. The patient is required to rate each item in a 5-point scale, ranging from 0 (very little) to 4 (very much). The ASI has adequate test/retest reliability.
Fear Questionnaire (FQ) | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The FQ is a 15-item questionnaire that yields four scores: main phobia, global phobia, total phobia and anxiety-depression; the total phobia score is composed of agoraphobia, social and blood-injury subgroups. It is reliable and valid.
Social Interaction Anxiety Inventory (SIAS) | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The SIAS assesses fears of general social interaction. It comprises 20 items, rated on a 5-point Likert scale, from 0 (not at all characteristic of me) to 4 (extremely characteristic of me). Internal consistency and test-retest reliability is high.
Fear of negative evaluation scale | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The FNE is a 30-item true-false inventory measuring anticipation of and distress about being negatively evaluated by others.
Social avoidance and distress scale | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The SAD is a 28-item true-false questionnaire measuring subjective distress experienced in social situations and avoidance of such situations.
Panic Disorder Severity Scale (PDSS-SR) | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The PDSS-SR is a self-report that consists of seven items rating frequency of panic attacks on a 5-point scale from 0 to 4, being the total score 28. It has good test-retest reliability and is sensitive to change with treatment.
Agoraphobia Inventory | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  This instrument measures the types of altered responses (motor (to places, means of transportation, and situations), subjective psychophysiological, and cognitive) of the patient, alone and in company, to the most common stimulus situations, as well as the variability of altered responses. Among the proposed items, patients must also indicate the symptoms that cause them the most difficulties in daily life.
Overall Depression Severity and Impairment Scale | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The ODSIS is a five-item instrument designed to measure severity and impairment of depressive symptoms. Items are coded from 0 to 4 and are summed to obtain one total score.
Overall Anxiety Severity and Impairment Scale | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The OASIS is a five-item continuous measure of anxiety-related severity and impairment. Items are coded from 0 to 4 and are summed to obtain one total score. The OASIS have shown high internal consistency, excellent test-retest reliability, and convergent and discriminant validity in clinical and non-clinical samples (i.e., Norman et al., 2006)
Behavioral Avoidance Test | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  Behavioral Avoidance Tests (BATs) are fundamental tools in the assessment and treatment of specific anxiety disorders, such as claustrophobia, acrophobia, panic disorder, and social anxiety. For claustrophobia, a BAT may involve progressively entering confined spaces, such as an elevator or a windowless room, while recording their anxiety level and avoidance behavior. For acrophobia, a BAT could involve gradually climbing to elevated locations, such as stairs or balconies, allowing observation of how they tolerate exposure to height. For panic disorder, interoceptive BATs are used, in which feared physical sensations (such as hyperventilating or spinning in a chair) are induced to assess the patient's reaction to bodily symptoms associated with panic. On the other hand, in social anxiety, a common task in a BAT is to ask the patient to give a speech in front of a small audience or a camera, thereby assessing their level of discomfort, physiological arousal, and avoidance behaviors.

OTHER OUTCOMES:
DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) | Baseline, up to 12 weeks (average)
  DSM-5 criteria will be considered
The Clinician Severity Scale | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  It uses a scale from 0 (absent/none) to 8 (very disturbing/disabling).
Item Short Form Health Survey (SF-12) | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  The SF-12 is a self-report that measures the impact of health on everyday life. It comprises 12 items and it is a valid and reliable measure. The internal consistency is great.
Quality of Life Inventory | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  It is a 10-item self-report that assesses various aspects of quality of life. These dimensions are rated on a 10-point Likert scale, ranging from 1 (poor) to 10 (excellent). The dimensions include physical well-being, psychological/emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social-emotional support, community and services support, personal fulfillment, spiritual fulfillment, and overall perception of quality of life. The total score is calculated as the average of all items and ranges from 1 to 10, with scores between 1 and 4.5 indicating a perception of quality of life below average, scores between 4.6 and 8.1 indicating an average perception, and scores between 8.2 and 10 indicating a perception above average. Test-retest reliability (0.89) and internal consistency (α = 0.89) are strong; discriminant validity is demonstrated in a sample of patients with mental illness.
Patient's Improvement Scale (adapted from the Clinical Global Impression scale, CGI) | Baseline, up to 12 weeks (average), follow-ups (3 months, 6 months, 12 months)
  This scale is intended to evaluate the patient's degree of progress over their initial state. The patient rates the items on a scale of 1 (much worse) to 7 (much better).
The Expectation of Treatment and Satisfaction with the Treatment scale (adapted from Borkovec and Nau) | Baseline, up to 12 weeks (average)
  These two scales consist of six items each. Participants rate these items on a scale from 0 (strongly disagree) to 10 (strongly agree). Their aim is to evaluate the treatment's ability to meet the patients' expectations, its perceived logic, its potential for treating other psychological issues, its usefulness for the patient, the likelihood of recommending it to others and its aversion. The Expectation of Treatment Scale is completed after the description of the intervention, before receiving any treatment and the Satisfaction with the Treatment Scale is completed after it is finished, assessing the patient´s satisfaction with the intervention.
Qualitative Interview | Up to 12 weeks (average)
  A semi-structured interview developed ad-hoc based on the Expectation and Satisfaction Scale (adapted from Borkovec & Nau) following the principles specified in the CQR guidelines (Hill et al., 2005). This included different open-ended questions that assess satisfaction using the Exposure Therapy App; why they would recommend it to other people with ADs; utility; intrusiveness due to aspects of threat to confidentiality when using this technology; aspects of the tool that make it easier and/or more difficult to use.
Preferences Questionnaire | Up to 12 weeks (average)
  The Preference Questionnaire: Traditional In-Live Exposure vs. SYMPTOMS-JIT Exposure is a specially designed instrument to compare the acceptance of two exposure treatment modalities in people with anxiety disorders: one guided by a therapist in real-life settings and the other assisted by a mobile app that allows for autonomous task completion. Through ten items, the questionnaire assesses the patient's willingness to repeat each type of treatment, their preference, perceptions of efficacy, usefulness, logic, aversiveness, and recommendation to others, combining rating scales and multiple-choice options to obtain useful information in clinical or research contexts.
The System Usability Scale (SUS) | Baseline, up to 12 weeks (average)
  This scale is one of the most popular methods for assessing the usability of ICT applications. The concept of usability describes how simple it is for the users to use a technological tool to accomplish a certain task in a given situation. They must indicate how much they agree or disagree with the 10 items using a 5-point Likert scale, 1 being strongly disagree and 5 being strongly agree).
User Version of the Mobile Application Rating Scale | Up to 12 weeks (average)
  uMARS consists of 20 items assessing objective and subjective app quality, rated on a 5-point Likert scale ranging from 1 ("poor") to 5 ("excellent"). In addition, items 13-16 include the additional option of "not applicable." The objective quality score is calculated as the mean of the scores of 4 dimensions: engagement (items 1-5), functionality (items 6-9), esthetics (items 10-12), and information (items 13-16). A subjective quality score is obtained as the mean of 4 subjective items (17-20). The final uMARS subscale includes 6 items, designed to assess the perceived impact of the app on the user's awareness, knowledge, attitudes, intention to change, helpseeking, and the probability of changing the target health behavior, also rated on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree").

CONTACTS AND LOCATIONS:
Overall Officials: Juana María Bretón-López, Lecturer, Principal Investigator — University Jaume I; Carlos Granell, Lecturer, Principal Investigator — University Jaume I; Sven Casteleyn, Lecturer, Principal Investigator — University Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Plaisier I, Beekman AT, de Graaf R, Smit JH, van Dyck R, Penninx BW. Work functioning in persons with depressive and anxiety disorders: the role of specific psychopathological characteristics. J Affect Disord. 2010 Sep;125(1-3):198-206. doi: 10.1016/j.jad.2010.01.072. Epub 2010 Feb 24. PMID 20185180
- [Background] Miralles I, Granell C, Diaz-Sanahuja L, Van Woensel W, Breton-Lopez J, Mira A, Castilla D, Casteleyn S. Smartphone Apps for the Treatment of Mental Disorders: Systematic Review. JMIR Mhealth Uhealth. 2020 Apr 2;8(4):e14897. doi: 10.2196/14897. PMID 32238332
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- See also: Related Info — https://symptoms-app.com/index.html